CLINICAL TRIAL: NCT04857723
Title: Adaptation To and Satisfaction With Contact Lens Wear In Myopic Young Adults
Status: Completed | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-20-48
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2022-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Daily disposable contact lens (Experimental): Participants wore a daily disposable contact lens for 3 months.
  Interventions: Device: daily disposable contact lens

INTERVENTIONS:
Device: daily disposable contact lens — Daily disposable contact lens for 3 months

SUMMARY:
The purpose of this study was to assess whether young adults could adapt to and achieve satisfaction with a daily disposable contact lens.

DETAILED DESCRIPTION:
This was a prospective, single group, dispensing clinical trial to determine subjective and objective visual performance measures, patient satisfaction and adaptability to a commercially available daily disposable contact lens in myopic young adults over 3 months of daily lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Is between 17 and 25 years of age (inclusive) and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Has a vertex corrected spherical equivalent distance refraction that ranges between - 0.75D to -6.00D in each eye;
* Has astigmatism ≤ -0.75 DC in either eye, by refraction;
* Be correctable to better than 0.20 logMAR in each eye by refraction;
* Has habitually worn spherical soft contact lenses to correct for distance vision (i.e. no multifocal or monovision) for the past 3 months;
* Is willing to wear contact lenses for at least 10 hours a day, 6 days a week while in the study;
* Demonstrates an acceptable fit with the study lenses;
* Has ocular health findings considered to be "normal" and which would not prevent the participant from safely wearing contact lenses.

Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Has a history of amblyopia;
* Has TNO Stereoacuity worse than 120" arc / or Titmus worse than 100" arc;
* Has any known active ocular disease and/or infection;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
* Has known sensitivity to the diagnostic pharmaceutical (sodium fluorescein) to be used in the study;
* Is pregnant, lactating or planning a pregnancy at the time of enrolment (verbal confirmation at the screening visit);
* Is pseudophakic;
* Has undergone refractive error surgery;
* Has one of following experiences with MiSight lenses:
* Is currently wearing MiSight lenses or
* Has worn MiSight lenses for more than one week at any given time or
* Has worn MiSight lenses for any more than 30 minutes in the past 30 days;
* Has had orthokeratology treatment within the last 3 months.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily Disposable Contact Lens
Started | 29
Completed | 27
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Twenty-nine participants enrolled in the study and 27 completed the study. Demographic information was recorded for the 2 discontinued patients and therefore included in the baseline population.
Arm/Group | Daily Disposable Contact Lens
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Quality of Vision (QoV)
Description: The Subjective Quality of Vision (QoV) questionnaire consisted of 30 items assessing 10 visual symptoms. Each symptom was evaluated using three sub-questions: frequency, severity, and bothersomeness. All subquestions were rated on a 4-point scale from 0 to 3, where higher values represent a higher severity, frequency, or bothersomeness. For analysis, each dimension-frequency, severity, and bothersomeness-was treated independently. Scores for each were calculated by summing the responses across all 10 symptoms, resulting in separate total scores for each dimension. Each total score ranged from 0 to 30. Thus, the Overall Frequency of Symptoms, Overall Severity, and Overall Bothersomeness scores each represent the sum of the respective ratings across all visual symptoms.
Time Frame: 3 months
Population: The 2 discontinuations occurred after lens dispensing but prior to the first follow up visit. These participants were excluded from the data analysis population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily Disposable Contact Lens
Number analyzed (Participants) | 27
score on a scale
  Overall Frequency | 6.1 (3.6)
  Overall Severity | 5.3 (3.5)
  Overall Bothersomeness | 4.7 (4.1)

2. Secondary Outcome: Contact Lens Impact on Quality of Life (CLIQ)
Description: Participant quality of life was measured after 3 months of lens wear using a CLIQ 28-item questionnaire. Each question was scored on a 1-5 integer scale, where 1=never and 5=always. As written, scores were not consistently associated with a better or worse outcome. An algorithm was later applied for consistency (i.e., for categories [1,2,3,4,5], for the first 20 questions [5,4,3,3,3] are assigned and for 21-28 [2,2,3,4,5]). After the conversion, the average of all scores was used to measure the CLIQ. The CLIQ score ranged from a minimum of 2.71 to a maximum of 5, with 5 representing the best score.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily Disposable Contact Lens
Number analyzed (Participants) | 27
score on a scale | 4.1 (0.5)

ADVERSE EVENTS:
Time Frame: The duration of the study, approximately 3 months.
Arm/Group | Daily Disposable Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 4/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Disposable Contact Lens (N=27)
Corneal infiltrates (Eye disorders) | 1 (1)
Burn (General disorders) | 1 (1) — Burns on leg due to spilled drink. Unrelated to lens.
Corneal staining (Eye disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT04857723/Prot_SAP_000.pdf